CLINICAL TRIAL: NCT02721563
Title: A Perspective Random Trial of Sodium Glycididazole Combined With Definitive Concurrent Chemoradiotherapy for Locally Advanced Squamous Cell Esophageal Carcinoma
Brief Title: A Trial of CMNa Combined With Definitive Concurrent Chemoradiotherapy for Locally Advanced ESCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, president, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMNAER2
Record Dates: First submitted 2016-03-09; First posted 2016-03-29 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — sodium glycididazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Glycididazole (Active Comparator): Sodium Glycididazole：800mg/m2，finished in 30 minutes,within 60 minutes after intravenous drip for radiation therapy.Three times a week (once every other one day),before radiation therapy. Chemotherapy Paclitaxel:45 mg/m²,d1,week 1-6 Cisplatin:20 mg/m²,d1,week 1-6 OR Docetaxel: 75 mg / m², 1 day or divided into D1, D8 days, 21 days / cycle. Cisplatin: 75 mg / m², divided into D1-D3 days or D1-D5 days, 21 days / cycle. Or nedaplatin: 80 mg / m², 21 days / cycle.
  OR 5-FU: 500 mg / m² / day, divided into D1 ~ D5 for use, 21 days / cycle. Cisplatin: 75 mg / m² / day, divided into D1-D3 day or D1-D5 days, 21 days / cycle. Or nedaplatin: 80 mg / m², 21 days / cycle 3DCRT/IMRT:2.0Gy/f/day,T60Gy/30f,week 1-6
  Interventions: Drug: Sodium Glycididazole
- Control Group (Placebo Comparator): Placebo：dissolved in 100mlphysiological saline(Now with chef),ivgtt,finished in 30 minutes,within 60 minutes after intravenous drip for radiation therapy.Three times a week (once every other one day),before radiation therapy, total 6 weeks course.Chemotherapy Paclitaxel:45 mg/m²,d1,week 1-6 Cisplatin:20 mg/m²,d1,week 1-6 OR Docetaxel: 75 mg / m², 1 day or divided into D1, D8 days, 21 days / cycle. Cisplatin: 75 mg / m², divided into D1-D3 days or D1-D5 days, 21 days / cycle. Or nedaplatin: 80 mg / m², 21 days / cycle.
  OR 5-FU: 500 mg / m² / day, divided into D1 ~ D5, 21 days / cycle. Cisplatin: 75 mg / m² / day, divided into D1-D3 day or D1-D5 days, 21 days / cycle. Or nedaplatin: 80 mg / m², 21 days / cycle 3DCRT/IMRT:2.0Gy/f/day,T60Gy/30f,week 1-6
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Glycididazole — Sodium Glycididazole 700mg/m2.Three times a week (once every other one day),before radiation therapy, total 6 weeks.
  Arms: Sodium Glycididazole
Drug: Placebo — Placebo:three times a week (once every other one day),before radiation therapy, total 6 weeks.
  Arms: Control Group

SUMMARY:
This is a perspective, multicenter,randomized controlled trial to evaluate the efficacy and safety of treatment with CMNa combined with concurrent chemoradiotherapy in patients with locally advanced squamous cell esophageal carcinoma . Analyses of primary objective (ORR) will be done as defined in the protocol.

DETAILED DESCRIPTION:
The primary end point of this study is objective response rate.The secondary end point is OS, PFS and the safty of drug. The primary hypothesis is the CMNa will improve ORR and thus improve OS, PFS. Assuming bilateral a=0.05, statistical power of 80%.The total sample size is 104 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to study entry
2. Patients with ESCC in upper and middle thoracic segment（stage II-III）confirmed by imaging and pathology or cytology, which is unsuitable or refuse surgery;
3. Capable for chemo-radiotherapy;
4. The existence of measurable lesions;
5. ECOG PS of 0 or 1
6. Possible semi-liquid diet;
7. Expected lifetime≥3 months
8. normal bone marrow reserve: ANCcount ≥1500/mm3;platelet count ≥100,000/ mm3,hemoglobin≥9g/dl
9. normal hepatic funcion:bilirubin level ≤1.5×ULN;AST/ALT≤1.5×ULN
10. normal renal function: serum creatinine≤1.5mg/dl and calculated creatinine clearance ≥60ml/min
11. normal cardiac function
12. Subjects tumor tissue available for the relevant biomarker detection

Exclusion Criteria:

1. Female subject who is during pregnancy or lactation, and the subject who have fertility don't take effective contraception during study
2. Any mental illness or nervous system lesions or can't tell treatment response clearly (such as cerebrovascular accident sequelae)
3. Any serious uncontrolled disease and infection, such as severe heart, liver, kidney diseases or diabetes, can't complete the treatment plan
4. Patients who have other malignant lesions, except curable skin cancer (non-melanoma skin cancer),carcinoma in situ of cervix or serve disease cured for 5 years
5. Primary lesions were multifocal
6. Patients who have obvious esophageal ulcers or have above moderate pains in chest-back or have symptoms of esophageal perforation
7. received anti-cancer treatment of esophageal cancer before the group, including surgery, radiotherapy, chemotherapy (induction of chemotherapy before the group is greater than or equal to two cycles).
8. Not esophageal squamous carcinoma confirmed by pathology or cytology
9. History of active hepatitis
10. Unable to comprehend the study requirement or who are not likely to comply with the study requirements
11. Significant disease which, in the investigator's opinion, would exclude the patient from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 3 months

SECONDARY OUTCOMES:
Overall survival | 36 months
Progression free survival | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, Ph.D, M.D, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (10):
- China (10):
  - Qianfoshan Hospital of Shandong, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - Jining NO.1 People's Hospital, Jining, Shandong
  - Liaocheng People 's Hospital, Liaocheng, Shandong
  - Qingdao Center Medical Group, Qingdao, Shandong
  - Rizhao City People 's Hospital, Rizhao, Shandong
  - Fei Cheng People's Hospital, Tai’an, Shandong
  - An Qiu People's Hospital, Weifang, Shandong
  - The Fourth People's Hospitalof Zibo, Zibo, Shandong

IPD SHARING:
Plan to Share IPD: No